CLINICAL TRIAL: NCT04704908
Title: Immuno-persistence Study of A Bivalent Human Papillomavirus (Type 16, 18) Recombinant Vaccine (E.Coli) in Healthy Female Subjects Aged 9 to 17 Years
Brief Title: Immuno-persistence Study of a Recombinant Human Papillomavirus 16/18 Bivalent Vaccine in Preadolescent Girls (54m)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jun Zhang (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jun Zhang, Professor, Xiamen University
Organization: Xiamen University (Other)
Other Study IDs: HPV-PRO-006-3
Record Dates: First submitted 2021-01-07; First posted 2021-01-12 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; Vaginal Intraepithelial Neoplasia; Vulvar Intraepithelial Neoplasia; Persistent Infection
Keywords: Human Papilloma Virus 16; Human Papilloma Virus 18; adolescent girl; non-inferiority; immuno-persistence
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Persistent Infection | interventions — Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 9-17y (0,1,6m): Participants in this arm have received 60μg of HPV 16/18 bivalent vaccine according to 3 doses of HPV 16/18 bivalent vaccine
  Interventions: Drug: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli)
- 9-14y (0,6m): Participants in this arm have received 60μg of HPV 16/18 bivalent vaccine according to 2 doses of HPV 16/18 bivalent vaccine
  Interventions: Drug: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli)
- 18-26y (0,1,6m): Participants in this arm have received 60μg of HPV 16/18 bivalent vaccine according to 3 doses of HPV 16/18 bivalent vaccine
  Interventions: Drug: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli)

INTERVENTIONS:
Drug: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) — The bivalent HPV-16/18 vaccine was a mixture of two aluminum hydroxide adjuvant-absorbed recombinant L1 VLPs of HPV-16 and HPV-18 expressed in E. coli. A 0.5 ml dose of the bivalent HPV test vaccine comprised 40 μg of HPV-16 and 20 μg of HPV-18 L1 VLPs absorbed with 208 μg of aluminum adjuvant
  Other Names: There is no other Intervention in this study

SUMMARY:
The primary objective of this study is to evaluate the immuno-persistence (type specific IgG antibody) of the tested vaccine administered in girls aged 9-17 years,comparing to young healthy adults of 18-26 years who received the standard 3-dose schedule (0,1,6 months).

DETAILED DESCRIPTION:
This is a follow-up study that is based on the bridging study of a recombinant human papillomavirus 16/18 bivalent vaccine in preadolescent girls(Unique Protocol ID:HPV-PRO-006,Identifiers: NCT02562508) .The investigators will recruit people who have participated in bridging study before and collect their serum samples to test the seroprevalence and geometric mean concentrations of anti-HPV16 and anti-HPV18 antibody on 54 months after dose 1

ELIGIBILITY:
Inclusion Criteria:

1. Participants who participated in the bridging study of a recombinant human papillomavirus 16/18 bivalent vaccine in preadolescent girls (Unique Protocol ID: HPV-PRO-006, Identifiers: NCT02562508) and received at least one dose;
2. Participants or participants and their legal guardians can fully understand the study content and sign an informed consent form；
3. Able to comply with the requests of the study;

Exclusion Criteria:

1. Participants with coagulation dysfunction (such as coagulation factor deficiency, blood-clotting disorder, or platelet disorder) or coagulation disorders, as diagnosed by a physician after vaccination ;
2. According to the investigator's judgment, there might be some medical, psychological, social or occupational factors which might impact on the individual to obey the protocol or sign the informed consent;
3. Abnormal blood clotting function or coagulopathy

Ages: 14 Years to 32 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Participants who participated in the bridging study (Unique Protocol ID: HPV-PRO-006, Identifiers: NCT02562508) and received at least one dose will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 979 (Estimated)
Dates: Start 2021-02-06 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Anti-HPV16 and anti-HPV18 seroprevalence and geometric mean concentrations at Month 54 (type-specific IgG antibody) | Month 54
  To detect the anti-HPV 16 and anti-HPV 18 type-specific IgG antibody level on 54 month after the dose 1

SECONDARY OUTCOMES:
Anti-HPV16 and anti-HPV18 seroprevalence and geometric mean concentrations at Month 54 (type specific neutralizing antibody) | Month 54
  To detect the anti-HPV 16 and anti-HPV 18 type specific neutralizing antibody level on 54 month after the dose 1

CONTACTS AND LOCATIONS:
Overall Officials: Ting Wu, Ph. D., Study Chair — Xiamen University
Locations (1):
- Jiangsu Provincial Centre for Disease Control and Prevention, Nanjing, Jiangsu, China